CLINICAL TRIAL: NCT06304740
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of a Single Subcutaneous Dose of IMG-007 in Healthy Participants
Brief Title: Safety and Pharmacokinetics of Subcutaneous Dose of IMG-007 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Cohorts 1 and 2 were completed. Cohort 3 was cancelled because it was no longer necessary based on information from another study. No safety concerns were noted.
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMG-007-102
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IMG-007 Cohort 1 (Healthy Participant) (Experimental): Cohort 1 will receive a single subcutaneous dose of IMG-007 Dose 1 or matching placebo.
  Interventions: Drug: IMG-007; Drug: Placebo
- IMG-007 Cohort 2 (Healthy Participant) (Experimental): Cohort 2 will receive a single subcutaneous dose of IMG-007 Dose 2 or matching placebo.
  Interventions: Drug: IMG-007; Drug: Placebo
- IMG-007 Cohort 3 (Healthy Participant) (Experimental): Cohort 3 will receive a single subcutaneous dose of IMG-007 Dose 3 or matching placebo.
  Interventions: Drug: IMG-007; Drug: Placebo

INTERVENTIONS:
Drug: IMG-007 — Subcutaneous injection of IMG-007
Drug: Placebo — Subcutaneous Injection of Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled study to assess the safety and PK profile of a single subcutaneous dose of IMG-007 in healthy participants. The study will comprise of a 5-week screening period, a 3-day In-patient Period in a clinical research unit (CRU) and an Out-patient Follow-up Period up to 127 days. The study will include 3 dose cohorts which will be enrolled sequentially. Participants will receive a single subcutaneous dose of IMG-007 or placebo at Baseline according to their assigned dose.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 18.0 kg/m2 and less than or equal to 32 kg/m2, and a minimum body weight of 50 kg for males and 45 kg for females
* Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.
* Female participants who are not pregnant or breastfeeding and meet at least one of the following conditions: not of childbearing potential or of childbearing potential and agrees to use a highly effective method of contraception.
* Male participants who agree to practice true abstinence or agree to use highly effective methods of contraception with female partners of childbearing potentials or are surgically sterilized.

Exclusion Criteria:

* Conditions or laboratory abnormality that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into the study.
* Major surgery ≤ 4 weeks before the Baseline Visit or planned major surgical procedure during the study.
* Use of any prescription medication (except for hormonal contraceptives for female participants within the 14 days prior to the first dose.
* Drug or alcohol abuse.
* Use of more than 5 tobacco/nicotine-containing products per month within 3 months of the first dose.
* Hepatitis B, hepatitis C, or human immunodeficiency virus infection.
* Evidence of latent tuberculosis (TB) or a history of untreated or inadequately treated TB infection.
* Receipt of a live/live attenuated vaccine within 2 months prior to Baseline Visit.
* Hypersensitivity to study treatment or other biologics
* Participation in prior IMG-007 study or another research study involving an investigational product within 30 days (small molecule) or 3 months (biological product), or 5 half-lives (whichever is longer) prior to the Baseline (Day 1) Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Adverse Event Evaluation | Up to 18 weeks
  Incidence of adverse events emergent from a single subcutaneous dose of IMG-007 in healthy participants.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters, Cmax | Up to 18 weeks
  Peak serum concentration following the administration of a single subcutaneous dose of IMG-007
Pharmacokinetic Parameters, Tmax | Up to 18 weeks
  Time to peak serum concentration following the administration of a single subcutaneous dose of IMG-007
Pharmacokinetic Parameters, AUC0-t | Up to 18 weeks
  Area under the concentration-time curve from time 0 until the last observed concentration following the administration of a single subcutaneous dose of IMG-007

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Australia

IPD SHARING:
Plan to Share IPD: Undecided